CLINICAL TRIAL: NCT02198495
Title: Continuous Versus Periodic Intravenous Iron Supplementation in Maintenance Hemodialysis Patients
Brief Title: Comparison Study of Two Iron Compounds for Treatment of Anemia in Hemodialysis Patients
Acronym: COPEFER
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gere Sunder-Plassmann, Prof. Dr., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COPEFER
Record Dates: First submitted 2014-07-18; First posted 2014-07-23 (Estimated); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: Anemia of Chronic Kidney Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ferric carboxymaltose (Active Comparator): Supplementation of ferric carboxymaltose 500 mg at week 0, 10, 20, 30
  Interventions: Drug: Supplementation of ferric carboxymaltose
- Iron sucrose (Active Comparator): Supplementation of iron sucrose 100 mg at week 0, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, 30, 32, 34, 36, 38
  Interventions: Drug: Supplementation of iron sucrose

INTERVENTIONS:
Drug: Supplementation of ferric carboxymaltose
  Arms: Ferric carboxymaltose
Drug: Supplementation of iron sucrose
  Arms: Iron sucrose

SUMMARY:
Patients with end-stage kidney disease on maintenance hemodialysis frequently require iron supplementation to compensate for ongoing iron losses, and to maintain hemoglobin levels with or without additional use of erythropoiesis-stimulating agents (ESA).

The investigators aim to compare two different intravenous iron preparations, ferric carboxymaltose and iron sucrose in 140 hemodialysis patients. The investigators primary objective is to assess whether both agents are equally effective to maintain a target haemoglobin within 10-12 mg/dl. The investigators will also measure ferritin, transferrin, transferrin saturation, and how much ESA therapy is administered.

Patients will be randomly assigned to either treatment group and followed in parallel over an active study period of 40 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Male and female patients aged ≥ 18
* Patients with anemia and end stage kidney disease on dialysis
* Hemoglobin ≥ 8,5g/dl
* Ferritin < 1000mg/dl
* TSAT < 50%
* CRP < 5mg/dl

Exclusion Criteria:

* Hemoglobin < 8,5g/dl
* Pregnancy or Nursing
* Known allergic reaction to i.v. iron supplementation or to ingredients of Investigational Medicinal Product (IMP)
* Chronic infections (HIV, Hep B, Hep C)
* Acute infections (CRP>5mg/dl; Antibiotic therapy except for prophylactic use)
* Malignant tumor disease
* Oral iron supplementation at study inclusion
* Participation in a different study at the same time
* Active bleeding issues
* Surgical intervention within the last 4 weeks before study inclusion
* Mental diseases
* Bronchial asthma
* Atopic allergy
* Eczema
* Receipt of red blood cell (RBC) concentrate within the last 4 weeks before study inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Serum hemoglobin level (g/dl) | 40 weeks

SECONDARY OUTCOMES:
Serum ferritin level (µg/l) | Week 0, 10, 20, 30, 40
Serum transferrin level (mg/dl) | Week 0, 10, 20, 30, 40
Serum level of transferrin saturation (TSAT) (%) | Week 0, 10, 20, 30, 40
ESA consumption in I.E./week or µg/week as appropriate | Week 0, 10, 20, 30, 40

CONTACTS AND LOCATIONS:
Overall Officials: Gere Sunder-Plassmann, MD, Principal Investigator — Medical University of Vienna
Locations (2):
- Austria (2):
  - Medical University of Vienna, Division of Nephrology and Dialysis, Vienna
  - Wiener Dialysezentrum GmbH, Vienna

REFERENCES:
- [Derived] Bielesz B, Lorenz M, Monteforte R, Prikoszovich T, Gabriel M, Wolzt M, Gleiss A, Horl WH, Sunder-Plassmann G. Comparison of Iron Dosing Strategies in Patients Undergoing Long-Term Hemodialysis: A Randomized Controlled Trial. Clin J Am Soc Nephrol. 2021 Oct;16(10):1512-1521. doi: 10.2215/CJN.03850321. Epub 2021 Sep 1. PMID 34470831